CLINICAL TRIAL: NCT03446352
Title: Multimodal Exercise Programs for Fall Prevention - Psychomotor Versus Psychomotor Combined With Whole-Body Vibration: A Randomized Controlled Trial
Brief Title: Multimodal Exercise Programs for Fall Prevention: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Collaborators: São João de Deus School of Nursing (Unknown); Horizon 2020 - Portugal 2020 (ALT20-03-0145-FEDER-000007 - Project: ESACA) (Unknown)
Responsible Party: Principal Investigator, Hugo Filipe Zurzica Rosado, MSc, University of Évora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UEvora
Record Dates: First submitted 2018-02-07; First posted 2018-02-26 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Fallers; High Risk of Falling
Keywords: Falls; Elderly; Psychomotor exercise program; Whole body vibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psychomotor exercise program (Experimental): The experimental group 1 (EG1) intervention comprises a psychomotor program. The program integrates 3 sessions / week of 75 minutes on alternated days. The psychomotor intervention includes exercises promoting simultaneous motor and cognitive stimulation (interval training).
  Interventions: Other: Psychomotor exercise program
- Combined exercise program (Experimental): The experimental group 2 (EG2) intervention combines the psychomotor program with a WBV program. The program integrates 3 sessions / week of 75 minutes (including the 6 minutes of WBV) on alternated days.
  Interventions: Other: Combined exercise program
- Control Group (No Intervention): Usual care. After the study, control group (CG) participants will be offered the opportunity to integrate a similar fall prevention program.

INTERVENTIONS:
Other: Psychomotor exercise program — Each session includes: beginning ritual (5 min), warm-up (15 min), main section comprising the multimodal exercises (40 min), cool-down (10 min), and finishing ritual (5 min).
  At the initial stage, the activation of different muscle groups will be performed, providing an elevation of the neurophysiological parameters. The main section (multimodal exercises) will be focused on the specific objectives through sensorimotor and neurocognitive activities. This section includes periods ranging 10-15 min of exercises mainly focused on motor stimulation- physical performance (cardiovascular, strength, balance, flexibility, agility and movement accuracy)- alternating with exercises mainly focused on cognitive stimulation- executive functions (planning ability, information processing speed, attention and dual-task performance).
  At the cool-down the participants will normalize their physiological parameters. Finally, at the finishing ritual the participants share their sensations experienced.
  Arms: Psychomotor exercise program
Other: Combined exercise program — The EG2 intervention combines the psychomotor exercise program with a WBV program. The program integrates 3 sessions / week of 75 minutes (including the 6 minutes of WBV) on alternated days.
  The WBV will integrate 3 sessions / week of 6 minutes each, with programed increased exercise time, series, and frequencies throughout the intervention.
  Arms: Combined exercise program

SUMMARY:
The aim of present study is to analyze and compare the effect of two exercise programs - psychomotor exercise program vs exercise combined program (psychomotor + whole body vibration) - on risk factors for falls of community-dwelling older adults who are fallers or are "at high risk of falling".

This experimental study is a randomized controlled trial. The program will run for 24 weeks (3 sessions / week of 75 minutes), followed by 12 weeks of follow-up without intervention. Participants of the groups will be assessed 1) at baseline, 2) at 12 weeks, 3) at 24 weeks, and 4) after the follow-up. Participants will be randomly allocated to three groups: experimental group 1 (psychomotor program); experimental group 2 (combined program) and control group.

DETAILED DESCRIPTION:
Aging is associated with a decline in executive functions, negatively influencing the motor, social and emotional capacities of older adults. (1) These losses will contribute to increase the risk of falling, so much that most falls occur during the performance of a dual-task (DT) (2).

The lack of balance, strength and poor body composition are seen as causes of falls, and should therefore be considered in the prevention programs of these events in older adults. (3-5) A psychomotor exercise program uses the body and movement as mediators, relying on the prevention of cognitive, sensory, perceptive, emotional and affective deterioration, exploring the neuroplasticity. (6,7) Therefore, this sensorimotor and neurocognitive program may prevent falls, but it is important to analyze its real impact in reducing either falls or the risk factors for falls in the older adults. No studies focusing on this subject were found.

The intervention through the whole body vibration (WBV) is referred in the literature as promoting the improvement of balance, mobility and agility, and preventing falls in the older adults.(8,9) WBV will have long-term therapeutic effects promoting the increase of muscle strength and increased bone mineral density. (10) Being two intervention methods with potential good results on falls prevention, it is not known whether there will be additional benefits in an intervention that combines both methods.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥65 years;
* Community-dwelling older adults;
* Older adults who have fallen in the last 6 months or who are at high risk of falling (scoring ≤25 points on Fullerton Advanced Balance Scale);
* Participation agreement;

Exclusion Criteria:

* Presence of severe cognitive decline (patients with a Mini-Mental State Examination ≤9);
* Fracture in one or both lower limbs for less than 4 months;
* Diagnosed of health conditions compromising the program participation, such as: severe osteoporosis (T ≤ 2.5, with the occurrence of one or more associated osteoporotic fractures); hip or knee prostheses; incapacitating cardiovascular conditions; epilepsy; cancer or metastases;
* Do not wish to participate in the study;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline, between and within groups comparison, in Executive Function | 0,3,6,9 months
  Outcome Measure - Trial Making Test (Part A and B) to assess information processing speed
Change from Baseline, between and within groups comparison, in Executive Function | 0,3,6,9 months
  Outcome Measure - Deary-Liewald Reaction Timed task to assess single and dual-task performance
Change from Baseline, between and within groups comparison, in Executive Function | 0,3,6,9 months
  Outcome Measure - Timed Up and Go (dual-task version) to assess dual-task performance
Change from Baseline, between and within groups comparison, in Executive Function | 0,3,6,9 months
  Outcome Measure - The d2 Test of Attention to assess attention
Change from Baseline, between and within groups comparison, in Physical Performance | 0,3,6,9 months
  Outcome Measure - Biodex (Peak Torque) to assess lower-body strength
Change from Baseline, between and within groups comparison, in Physical Performance | 0,3,6,9 months
  Outcome Measure - Senior Fitness Test (30-s Chair Stand Test) to assess lower-body strength
Change from Baseline, between and within groups comparison, in Physical Performance | 0,3,6,9 months
  Outcome Measure - Timed Up and Go (single and dual-task version) to assess agility
Change from Baseline, between and within groups comparison, in Physical Performance | 0,3,6,9 months
  Outcome Measure - Static Posturography Platform to assess balance
Change from Baseline, between and within groups comparison, in Physical Performance | 0,3,6,9 months
  Outcome Measure - Fullerton Advanced Balance Scale, ranging from 0 (worst) to 40 (best) points, to assess balance
Change from Baseline, between and within groups comparison, in Body Composition | 0,3,6,9 months
  Outcome Measure - Dual-energy X-ray Absorptiometry to assess body fat mass (%) and body lean mass (%)
Change from Baseline, between and within groups comparison, in Body Composition | 0,3,6,9 months
  Outcome Measure - Dual-energy X-ray Absorptiometry to assess bone mineral density
Fall occurrence in the previous 6 months at baseline and at post-intervention | 0,6 months
  Comparasion of the number of falls between and within groups

SECONDARY OUTCOMES:
Borg Rating of Perceived Exertion | 0-6 months
  Exercise intensity
Mini-Mental State Examination | 0 months
  Cognitive state
Composite Physical Function scale | 0 months
  Physical independence
International Physical Activity Questionnaire | 0 months
  Physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade de Évora, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bherer L. Cognitive plasticity in older adults: effects of cognitive training and physical exercise. Ann N Y Acad Sci. 2015 Mar;1337:1-6. doi: 10.1111/nyas.12682. PMID 25773610
- [Background] Lima LC, Ansai JH, Andrade LP, Takahashi AC. The relationship between dual-task and cognitive performance among elderly participants who exercise regularly. Braz J Phys Ther. 2015 Mar-Apr;19(2):159-66. doi: 10.1590/bjpt-rbf.2014.0082. Epub 2015 Apr 27. PMID 25993629
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] World Health Organization. Falls. [online]. 2016; Avaliable at: http://www.who.int/mediacentre/factsheets/fs344/en/
- [Background] Latorre Roman PA, Garcia-Pinillos F, Huertas Herrador JA, Cozar Barba M, Munoz Jimenez M. Relationship between sex, body composition, gait speed and body satisfaction in elderly people. Nutr Hosp. 2014 Oct 1;30(4):851-7. doi: 10.3305/nh.2014.30.4.7669. PMID 25335673
- [Background] Oliveira V, Carvalho S, Cardoso T. (2015). Quando o envelhecimento acontece. Rio de Janeiro: Wak Editora. Atualidades da Prática Psicomotora. 2015; 217-233.
- [Background] Fernandes, J. A Gerontopsicomotricidade como Práxis Terapêutica de Mediação Corporal. Journal of Aging and Innovation. 2014; 3 (3).
- [Background] Smith DT, Judge S, Malone A, Moynes RC, Conviser J, Skinner JS. Effects of bioDensity Training and Power Plate Whole-Body Vibration on Strength, Balance, and Functional Independence in Older Adults. J Aging Phys Act. 2016 Jan;24(1):139-48. doi: 10.1123/japa.2015-0057. Epub 2015 Jul 23. PMID 26215362
- [Background] Orr R. The effect of whole body vibration exposure on balance and functional mobility in older adults: a systematic review and meta-analysis. Maturitas. 2015 Apr;80(4):342-58. doi: 10.1016/j.maturitas.2014.12.020. Epub 2015 Jan 12. PMID 25631348
- [Background] Rauch F. Vibration therapy. Dev Med Child Neurol. 2009 Oct;51 Suppl 4:166-8. doi: 10.1111/j.1469-8749.2009.03418.x. PMID 19740225
- [Derived] Rosado H, Bravo J, Raimundo A, Carvalho J, Pereira C. Optimizing Cognitive and Physical Gains in Older Adults: Benefits of a Psychomotor Intervention Program Based on Functional Level. Medicina (Kaunas). 2025 Sep 2;61(9):1584. doi: 10.3390/medicina61091584. PMID 41010975
- [Derived] Rosado H, Bravo J, Raimundo A, Carvalho J, Almeida G, Pereira C. Can two multimodal psychomotor exercise programs improve attention, affordance perception, and balance in community dwellings at risk of falling? A randomized controlled trial. BMC Public Health. 2022 Jul 11;21(Suppl 2):2336. doi: 10.1186/s12889-022-13725-5. PMID 35818044
- [Derived] Rosado H, Bravo J, Raimundo A, Carvalho J, Marmeleira J, Pereira C. Effects of two 24-week multimodal exercise programs on reaction time, mobility, and dual-task performance in community-dwelling older adults at risk of falling: a randomized controlled trial. BMC Public Health. 2021 Nov 10;21(Suppl 2):408. doi: 10.1186/s12889-021-10448-x. PMID 34758759